CLINICAL TRIAL: NCT04886843
Title: The Effects Of Cold Application To The Intact Side In Addition Cross Training With NMES On Dorsiflexor Muscle Strength In Hemiplegia
Brief Title: Cold Therapy and Cross-Education of Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulPMRTRH-ct
Record Dates: First submitted 2021-05-09; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Cerebrovascular Stroke; Muscle Weakness
Keywords: Cold therapy; Cross-education; Neuromuscular electrical stimulation; Hemiplegia
MeSH Terms: conditions — Stroke; Muscle Weakness; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Therapy (Active Comparator): The patients have seated the knee joints in full extension and both ankle joints in a neutral position. Neuromuscular electrical stimulation (NMES) was applied to the non-affected side ankle dorsiflexors for five days, five sessions for a week. In addition to this application, a cold pack was applied on the affected side dorsiflexor muscle skin. The cold pack was applied on a moist towel for five minutes. A five-minute break was given and a further 5-minute cold application was repeated. The cold application was done simultaneously with NMES.
  Interventions: Other: Cold pack; Device: NMES
- Control (Placebo Comparator): The patients have seated the knee joints in full extension and both ankle joints in a neutral position. Neuromuscular electrical stimulation (NMES) was applied to the non-affected side ankle dorsiflexors for five days, five sessions for a week.
  Interventions: Device: NMES

INTERVENTIONS:
Other: Cold pack — Five minutes cold pack was applied on the affected side dorsiflexor muscle skin, a five-minute break was given and a further 5-minute cold application was repeated
  Arms: Cold Therapy
Device: NMES — NMES was applied to the nonaffected side ankle dorsiflexors

SUMMARY:
The aim of this study is to investigate whether a cold application to the contralateral (affected side) extremity in addition to unilateral neuromuscular electrical stimulation (NMES) application has a facilitating effect on muscle strength in post-stroke hemiplegia patients.

DETAILED DESCRIPTION:
In this prospective randomized controlled single-blind study, a total of 25 patients, 16 men, and 9 women were included according to inclusion and exclusion criteria. Patients were randomly assigned to the experimental group (n=12) or the control group (n=13). NMES has applied to the non-affected side ankle dorsiflexors five sessions for a week in both groups. In addition to the experimental group, the cold application was applied on the affected side dorsiflexor muscle skin. The cold application was done on a moist towel for five minutes using a cold pack. A five-minute break was given and a further 5-minute cold application was repeated. The cold application was done simultaneously with NMES. A conventional rehabilitation program was applied to all patients by a physiotherapist. Before and after treatment, both ankle dorsiflexor strength was measured with a force sensor. For force measurements, a force transducer (FC2211-0000-0100-L Compression Load Cell, TE Connectivity company, France) was used. Force transducer signals were received with a data acquisition device (POWERLAB® data acquisition system ADInstruments, Oxford, UK) and evaluated offline on the computer. The measurement values were expressed in kilogram.force (kg.f) and this value was normalized according to body weight.

ELIGIBILITY:
Inclusion Criteria:

* Cases with stroke duration ≥1 month
* Brunnstrom stage ≥4 for lower limb
* Unilateral stroke
* Ability to walk at least 10 m (FAC ≥3)
* Cooperating with the examination and tests

Exclusion Criteria:

* Cold allergy
* Active inflammatory, rheumatological, or infectious disease
* Presence of lower extremity fracture
* Severe spasticity (MAS> 3) in ankle dorsiflexors
* Peripheral nerve lesions such as polyneuropathy, radiculopathy
* Parent rhythm/conduction block problem in the heart
* Uncontrollable hypertension (Maxima >140 mmHg, Minima >90 mmHg)
* Have a contracture on the ankle joint
* The presence of skin lesions in the application area
* Finding or suspected active deep vein thrombosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change of ankle dorsiflexor isometric muscle strength | Change from Baseline ankle dorsiflexor isometric muscle strength at 6 days
  Force transducer used for measuring maximum voluntary ankle dorsiflexion force. The force unit is kilogram.force

SECONDARY OUTCOMES:
Change of Lower Extremity Brunnstrom Score | Change from Baseline Lower Extremity Brunnstrom Score at 6 days
  This test describes the sequences of motor recovery after stroke based on the muscle tone, synergy patterns and isolated movements. Brunnstrom classified stages of recovery into six stages. Stage 1 and 6. Stage 1:Flaccidity; Stage 6: Spasticity disappears and individual joint movements become possible
Change of Modified Ashworth Scale Score | Change from Baseline Modified Ashworth Scale Score at 6 days
  The modified Ashworth scale is the tool used to measure the increase of muscle tone. The modified Ashworth scale is score is graded between 0 and 4. 0: No increase in muscle tone, 4: Affected part(s) rigid in flexion or extension
Change of Functional Ambulation Scale Score | Change from Baseline Functional Ambulation Scale Score at 6 days
  The Functional Ambulation Classification (FAC) is a functional walking test that evaluates ambulation ability. Patients are categorized between 0 (non-functional ambulation) and 6 (independent).
Change of Timed Up and Go Test Score | Change from Baseline Change of Timed Up and Go Test Score at 6 days
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan Karacan, Assoc Prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sariyildiz M, Karacan I, Rezvani A, Ergin O, Cidem M. Cross-education of muscle strength: cross-training effects are not confined to untrained contralateral homologous muscle. Scand J Med Sci Sports. 2011 Dec;21(6):e359-64. doi: 10.1111/j.1600-0838.2011.01311.x. Epub 2011 Apr 18. PMID 21496110
- [Background] Lee M, Carroll TJ. Cross education: possible mechanisms for the contralateral effects of unilateral resistance training. Sports Med. 2007;37(1):1-14. doi: 10.2165/00007256-200737010-00001. PMID 17190532
- [Background] Howatson G, Zult T, Farthing JP, Zijdewind I, Hortobagyi T. Mirror training to augment cross-education during resistance training: a hypothesis. Front Hum Neurosci. 2013 Jul 24;7:396. doi: 10.3389/fnhum.2013.00396. eCollection 2013. PMID 23898251
- [Background] Ehrensberger M, Simpson D, Broderick P, Monaghan K. Cross-education of strength has a positive impact on post-stroke rehabilitation: a systematic literature review. Top Stroke Rehabil. 2016 Apr;23(2):126-35. doi: 10.1080/10749357.2015.1112062. Epub 2016 Feb 24. PMID 26907193
- [Background] Tokunaga T, Sugawara H, Tadano C, Muro M. Effect of stimulation of cold receptors with menthol on EMG activity of quadriceps muscle during low load contraction. Somatosens Mot Res. 2017 Jun;34(2):85-91. doi: 10.1080/08990220.2017.1299004. Epub 2017 Mar 21. PMID 28325123
- [Background] Shimose R, Ushigome N, Tadano C, Sugawara H, Yona M, Matsunaga A, Muro M. Increase in rate of force development with skin cooling during isometric knee extension. J Electromyogr Kinesiol. 2014 Dec;24(6):895-901. doi: 10.1016/j.jelekin.2014.08.002. Epub 2014 Aug 24. PMID 25218791